CLINICAL TRIAL: NCT03711838
Title: The Effect of Redox Potential on the Regulation of Satellite Cells and Skeletal Muscle Healing Following Exercise-Induced Muscle Damage
Brief Title: Redox Regulation of Satellite Cells and Skeletal Muscle Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Satellite Cells - UTH
Record Dates: First submitted 2018-10-11; First posted 2018-10-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Satellite Cells; Redox Status; Exercise-induced Muscle Trauma; Aseptic Inflammation
Keywords: Pax7; MyoD; Antioxidants; Myogenic potential; Skeletal muscle healing
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-Acetylcysteine (Experimental): N-Acetylcysteine supplementation: Orally, 40 mg/kg per day in 3 doses (250 ml each) for 7 consecutive days and immediately post-exercise. The remaining 8 days, 40mg/kg per day in 3 doses (250 ml each).
  Interventions: Dietary Supplement: N-Acetylcysteine
- Placebo (Active Comparator): Placebo administration: Orally 750 ml per day in 3 doses (250 ml each) for 7 consecutive days and immediately post-exercise. The remaining 8 days, 750 ml per day in 3 doses (250 ml each).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: N-Acetylcysteine — N-Acetylcysteine in a powder form diluted in a 250 ml drink containing 248 ml water and 2 ml of natural, non-caloric, flavoring-sweetener containing sucralose.
  Arms: N-Acetylcysteine
Dietary Supplement: Placebo — Placebo consisted of 248 ml water and 2 ml of natural, non-caloric, flavoring-sweetener containing sucralose.
  Arms: Placebo

SUMMARY:
Skeletal muscle stem cells (Satellite cells) are indispensable for muscle growth and remodeling following myofibril damage. Skeletal muscle trauma is present in numerous catabolic conditions, characterized by elevated proteolysis and muscle wasting such as, cancer cachexia and muscular dystrophy, which result in physical capacity impairment and a deteriorated quality of life. Recent studies performed in animals and cell cultures indicate that the increased levels of inflammation and oxidative stress and the reduction of antioxidant defense may blunt the satellite cells response and myogenic programming during muscle healing. However, evidence regarding the effects of redox status on satellite cells and muscle myogenic potential in humans is lacking. Exercise-induced muscle damage bears striking similarities with the aforementioned conditions, which makes it a valuable tool to investigate the redox-dependent regulation of satellite cells during muscle healing. Thus, the objectives of the present study are to examine the effects of redox status perturbation (via N-acetylcysteine administration) on intracellular pathways responsible for satellite cells responses at rest and following aseptic muscle trauma induced by damaging exercise.

DETAILED DESCRIPTION:
A total number of 40-60 young males aged 18-30 will be initially enrolled in the study. Then, participants will be allocated to either a 1) Low glutathione (GSH-low) or a 2) High glutathione (GSH-high) group based on the basal glutathione levels of their vastus lateralis muscle. In a double-blind, crossover, repeated measures design, participants will consume either Placebo (PLA) or N-acetylcysteine (NAC) before (7-day loading phase), on exercise day and for 8 consecutive days following a single bout of intense exercise (300 eccentric contractions at 30 deg/sec in an isokinetic dynamometer). In both conditions, blood samples and muscle biopsies will be collected at baseline, before the exercise protocol and at 2- and 8-days post-exercise. Muscle performance and soreness will also be assessed at the same time points. Before each trial, participants' dietary intake will be analyzed via diet recalls. Physical activity will be analyzed only at baseline via accelerometry. A 4-week washout period will be implemented between trials. Blood samples will be analyzed for inflammation and oxidative stress markers. Muscle samples will be analyzed for satellite cell responses and myogenic potential, protein levels of intracellular signaling proteins, muscle thiols and antioxidant enzyme activity.

ELIGIBILITY:
Inclusion Criteria:

1. No recent history of musculoskeletal injury
2. Non-smokers.
3. Abstain from any vigorous physical activity during the study
4. Abstain from consumption of caffeine, alcohol, performance-enhancing or antioxidant supplements, NSAIDs and medications before (at least 6 months) and during the study.

Exclusion Criteria:

1. A known NAC intolerance or allergy
2. A recent febrile illness
3. A recent history of muscle lesion and/or lower limb trauma
4. Presence of metabolic diseases
5. Use of anti-inflammatory medication.
6. Use of medication interacting with muscle metabolism.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in muscle satellite cells number (i.e. Pax7+ cells) and activation status (i.e. Pax7+/MyoD+ cells) | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Satellite cells number and activation status, will be assessed in muscle via immunohistochemistry.
Change in muscle myogenic mRNA expression | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  mRNA expression levels of Myogenic factor 5 (Myf5), myogenin and Myogenic factor 6 (Myf6/MRF4) and myostatin will be assessed in muscle using Real-Time Polymerase Chain Reaction (RT-PCR).
Change in muscle inflammatory state | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Pro-inflammatory (M1+) and anti-inflammatory (M2+) macrophages will be measured in muscle using immunohistochemistry.
Change in intracellular antioxidant enzymes in muscle | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Protein levels of Glutathione peroxidase 3 (GPx3), Superoxide dismutase 1 (SOD1) and Thioredoxin (Trx1) will be measured using western blotting.
Change in muscle thiol content | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration levels of reduced glutathione (GSH) and oxidized glutathione (GSSG) will be measured spectophotometrically.
Change in intracellular signaling proteins in muscle | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Protein levels of IGF-1, Notch1 and Wnt3 will be measured using western blotting.
Change in skeletal muscle damage levels | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Skeletal muscle damage will be quantified via histochemistry using H&E staining.

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) | At baseline
  RMR will be assessed after an overnight fast with participants in a supine position following a 15-min stabilization period by taking 30 consecutive 1-min VO2/CO2 measurements using a portable open-circuit indirect calorimeter with a ventilated hood system following a standard calibration protocol.
Body composition | At baseline
  Body composition will be measured using a dual-energy x-ray absorptiometry scanner (DXA).
Maximal oxygen consumption (VO2max) | At baseline
  VO2max will be assessed during continuous incremental running to volitional fatigue on a treadmill with a pulmonary gas exchange system (Oxycon Mobile; Sensor-Medics Corporation).
Isokinetic strength | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Maximal knee extensor eccentric peak torque at 60 degrees will be assessed on an isokinetic dynamometer.
Change in delayed onset of muscle soreness (DOMS) | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Muscle soreness will assessed during palpation of the muscle belly and the distal region of relaxed vastus medialis, vastus lateralis and rectus femoris following three repetitions of of a full squat. Subjects will rate their DOMS on a visual analogue scale (0-10).
Physical activity | At baseline.
  Level of habitual physical activity will be assessed using accelerometry (ActiGraph GT3X-BT accelerometer).
Dietary intake | At baseline.
  Daily dietary intake will be assessed using 7-day diet recalls.
Interleukin-1β (IL-1β) in blood | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of IL-1β will be measured in plasma.
Interleukin-6 (IL-6) in blood | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of IL-6 will be measured in plasma.
Interleukin-8 (IL-8) in blood | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of IL-6 will be measured in plasma.
Interleukin-10 (IL-10) in blood | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of IL-10 will be measured in plasma.
Cortisol in blood | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of cortisol will be measured in serum.
Protein carbonyls (PC) | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of protein carbonyls will be measured in muscle.
Malondialdehyde (MDA) | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of malondialdehyde will be measured in muscle.
Total antioxidant capacity (TAC) | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of TAC will be measured in serum.
Catalase | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of catalase will be measured in red blood cell lysate.
Creatine Kinase (CK) | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  Concentration of CK will be measured in serum.
White blood cell count in blood | At baseline, before the exercise protocol and at days 2 and 8 following exercise.
  White blood cell count will be measured in blood. White blood cell count will be measured in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Papanikolaou, PhD, Principal Investigator — University of Thessaly, School of Physical Education & Sport Science
Locations (1):
- Laboratory of Exercise Biochemistry, Exercise Physiology,and Sports Nutrition, School of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

REFERENCES:
- [Derived] Papanikolaou K, Jamurtas AZ, Poulios A, Tsimeas P, Draganidis D, Margaritelis NV, Baloyiannis I, Papadopoulos C, Sovatzidis A, Deli CK, Rosvoglou A, Georgakouli K, Tzatzakis T, Nikolaidis MG, Fatouros IG. Skeletal muscle and erythrocyte redox status is associated with dietary cysteine intake and physical fitness in healthy young physically active men. Eur J Nutr. 2023 Jun;62(4):1767-1782. doi: 10.1007/s00394-023-03102-2. Epub 2023 Feb 24. PMID 36828945
- [Derived] Papanikolaou K, Draganidis D, Chatzinikolaou A, Laschou VC, Georgakouli K, Tsimeas P, Batrakoulis A, Deli CK, Jamurtas AZ, Fatouros IG. The redox-dependent regulation of satellite cells following aseptic muscle trauma (SpEED): study protocol for a randomized controlled trial. Trials. 2019 Jul 31;20(1):469. doi: 10.1186/s13063-019-3557-3. PMID 31366396